CLINICAL TRIAL: NCT05796661
Title: Evaluation of Filters Useful Life, Metabolic Control, Electrolyte Profile and Acid-base Balance During Regional Anticoagulation With 4% Trisodium Citrate in Patients Undergoing CVVHDF: Effects of Increased Blood Flow
Brief Title: Patients Undergoing Continuous Venovenous Hemodiafiltration: Effects of Increased Blood Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRRT-QbTrial
Record Dates: First submitted 2023-03-14; First posted 2023-04-03 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury
Keywords: Continuous renal replacement therapy; Blood flow; Filtration fraction
MeSH Terms: conditions — Acute Kidney Injury | interventions — trisodium citrate

STUDY DESIGN:
Intervention Model Description: This is a randomized, crossover, single-center study, with inclusion of patients over a period of 11 months, between January 9, 2023 and November 30, 2023. We aim to include 27 patients. Randomized by raffle, which will be carried out manually in blocks divided into 3 envelopes numbered from 01 to 03, and within them will contain 9 papers, also numbered from 1 to 27 with the definition of control group and experimental group. Following the order from 01 to 03, the envelopes will have: envelope 1: 9 samples (5 for control group and 4 for experimental group); envelope 2: 9 samples (4 for control group and 5 for experimental group); envelope 3: 9 samples (5 for control group and 4 for experimental group). Groups: Qb150 (control group) (blood flow 150 mL/min), Qb250 (experimental group) (blood flow 250 mL/min). Time for each treatment: 72 hours. Crossover: after 72 hours. Treatment pause (wash-out): 4 (minimum) to 6 (maximum) hours.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qb150 (Experimental): This group will be exposed to continuous venovenous therapy with a blood flow of 150ml/min; already standardized by the institution; for a maximum time of 72 hours or interrupted sooner if the system clots or the filter loses patency.
  Both groups will have a "wash out" of 6 hours before crossing the arms of the work.
  Interventions: Other: Effects of increased blood flow during regional anticoagulation with 4% trisodium citrate in patients undergoing continuous venovenous hemodiafiltration
- Qb 250 (Active Comparator): This group will be exposed to continuous venovenous therapy with a blood flow of 250ml/min; experimental group to evaluate increased blood flow and filter durability; for a maximum time of 72 hours or interrupted sooner if the system clots or the filter loses patency.
  Both groups will have a "wash out" of 6 hours before crossing the arms of the work.
  Interventions: Other: Effects of increased blood flow during regional anticoagulation with 4% trisodium citrate in patients undergoing continuous venovenous hemodiafiltration

INTERVENTIONS:
Other: Effects of increased blood flow during regional anticoagulation with 4% trisodium citrate in patients undergoing continuous venovenous hemodiafiltration — Patients will be exposed to continuous venovenous renal therapy with distinct blood flows in 2 periods, to be defined by draw. The control group will have a flow of 150ml/min and the intervention group 250ml/min. Therapy is intended for a period of 72 hours (maximum defined by the manufacturer); with a 6-hour "washout" and, after that, the arm is changed to be exposed to the other blood flow.

SUMMARY:
Acute Kidney Injure (AKI) is a syndrome with high incidence and prevalence in Intensive Care Units (ICU). It is estimated that 50% of the in the sector present AKI at some point and 10 to 15% require renal replacement therapy (RRT). Although studies do not show the superiority of continuous methods, the most severely ill patients are directed to this type of RRT. A disadvantage of continuous therapies is the need for anticoagulation. Critically ill patients have a pro-clotting state (inflammation) and several risk factors for bleeding (coagulopathies, postoperative, large vessel puncture).

On the one hand, ineffective anticoagulation compromises the efficiency of the procedure, shortens the life of the extracorporeal system, consumes resources and increases blood loss due to unexpected and early filter clotting. There is no consensus on what would be the optimal blood flow (Qb) in continuous dialysis, especially when regional citrate anticoagulation (RCA) is used. Theoretically, a higher flow rate would prevent stasis in the system and decrease the risk of filter clotting. Studies show conflicting results. Increasing Qb from 150 to 250 mL/min showed that circuit life and the chance of coagulation were similar. On the other hand, blood flow is important for maintaining the filtration fraction (FF), the ratio of ultrafiltrate flow to plasma flow. Ideally, the FF should be kept below 25% to avoid hemoconcentration and coagulation of the filter. Therefore, the higher the convection rate, the higher the blood flow should be to keep the FF in the optimal range. Since the anticoagulation capacity of citrate is dependent on its concentration, around 4 mmol/L of blood, by increasing the blood flow, the citrate infusion is proportionally increased. Theoretically, the higher citrate load offered should be metabolized and, in theory, could cause its overload with the occurrence of metabolic alkalosis and hypernatremia. This situation occurs when its maximum metabolizing capacity is not reached and there is an excess of citrate infusion relative to the buffering requirement. Thus, we intend to evaluate filter useful life, metabolic control, electrolyte profile and acid-base balance in ICU patients undergoing continuous venovenous hemodiafiltration (CVVHDF), regional citrate anticoagulation during blood flow augmentation.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a clinical syndrome with a high incidence and prevalence in Intensive care units (ICU). It is estimated that 50% of ICU patients have AKI at some point.

About 10-15% of these individuals require renal replacement therapy (RRT). Although studies have not conclusively shown the superiority of continuous methods, the most severe patients are usually referred for this type of therapy.

The main indications for continuous therapies are hemodynamic instability, cardiogenic shock, severe respiratory insufficiency, risk situations for brain edema, hypercatabolism, need for strict volume control, acute liver disease and major sodium disturbances. One of the main disadvantages of continuous therapies is the necessity of anticoagulation. Critically ill patients have a pro-clotting state (inflammation) and several risk factors for bleeding (coagulopathies, postoperative, large vessel puncture). On the one hand, the lack or ineffective anticoagulation compromises the efficiency of the procedure, shortens the life of the extracorporeal system, consumes resources and increases blood loss due to unexpected and early filter coagulation. On the other hand, excessive use of anticoagulants, especially heparin, is associated with bleeding and increased transfusions.

In this scenario, regional anticoagulation with citrate (RCA) has become the method of choice in the different modalities of continuous dialysis. When compared to heparin, the use of regional citrate anticoagulation is associated with less bleeding and transfusion need and longer life of the extracorporeal system. It also seems to decrease endothelial activation, neutrophil degranulation and activation of the complement system.

The anticoagulate property of citrate is based on its binding to calcium (Ca). Citrate quenches Ca in the extracorporeal system, an essential cofactor in several steps of coagulation. Optimal anticoagulation is achieved when ionic Ca concentration in the extracorporeal circuit is maintained between 0.25 and 0.35 mmol/L. This is usually achieved with a citrate level in the circuit around 4mmol/L of blood. Depending on the modality chosen and other factors, up to 60% of the citrate-Ca complex is eliminated during passage through the filter (molecular weigh of 298 Daltons and partition coefficient of 1.0). The rest is metabolized in the Krebs cycle mainly in the liver, kidneys and skeletal muscles. Each mol of trisodium citrate causes 3 moles of bicarbonate thus correctly, partially or completely, the metabolic acidosis resulting from renal failure. Ca and sodium (Na) are released into the systemic circulation. Trisodium citrate also increases the strong ion difference due to the high sodium concentration in the solution, thus increasing the buffering capacity. In parallel it is necessary the Ca replacement to maintain normal calcemia. The citrate also quenches magnesium, which can lead to a disturbance of this electrolyte.

There is no consensus on what the optimal blood flow (Qb) would be in continuous dialysis, especially when using regional citrate anticoagulation. Theoretically, a higher blood flow would prevent stasis in the system and thus decrease the risk of filter coagulation. Studies show conflicting results. For example, one study evaluated increasing Qb from 150 to 250 mL/min and showed that circuit useful life and the chance of coagulation of the extracorporeal system were similar between the two groups. On the other hand, blood flow is important for maintaining the filtration fraction (FF), the ratio of ultra-filtrated flow to plasma flow (blood flow minus hematocrit). Ideally, the FF should be kept below 25% to avoid hemoconcentration and coagulation of the filter capillary fibers. So the higher the convection rate (ultrafiltration), the higher the blood flow should be to keep the FF in the optimal range.

Since the anticoagulation capacity of citrate is dependent on its concentration, around 4 mmol/L of blood, by increasing blood flow, citrate infusion is proportionally increased. Theoretically, the higher citrate load offered should be metabolized and, in theory, could lead to citrate overload with the occurrence of metabolic alkalosis and hypernatremia. This situation occurs when the maximum capacity of citrate metabolization is not reached and there is an excess of citrate infusion relative to the buffering requirement. The total Ca/systemic ionic Ca ration remains normal, below 2.5. The oversupply of citrate can be easily corrected by decreasing the bicarbonate concentration of the dialysate, increasing the dialysate dose or decreasing the citrate infusion.

Therefore, we intend to evaluate filter useful life, metabolic control, electrolyte profile and acid-base balance in ICU patients with AKI undergoing continuous venovenous hemodiafiltration (CVVHDF), regional anticoagulation with citrate during increased blood flow.

Hypothesis: Increasing blood flow during continuous venovenous hemodiafiltration prevents stasis in the system and thus reduces the risk of filter coagulation. Blood flow is important for maintaining the filtration fraction (FF), the ratio of ultrafiltrate flow to plasma flow (blood flow minus hematocrit). Ideally, the FF should be kept below 25% to avoid hemoconcentration and coagulation of the filter capillary fibers. So the higher convection rate (ultrafiltration), the higher the blood flow should be to keep the FF in the optimal range. Therefore, it is expected that higher blood flow (250 mL/min) will reduce the FF and concomitantly prolong the life of the filter.

ELIGIBILITY:
The inclusion criteria will be:

* Age greater than 18 years.
* Weight ≥ 50 Kg.
* Agreeing to participate in the study (TCLE duly elucidated and signed by the patient or family member/guardian).
* Admitted to the hospital ICU.
* Acute Kidney Injury in need of RRT and indication (according to the evaluation of the assistant nephrologist) of continuous therapy.

Exclusion criteria will be:

* Age < 18 years.
* Weight < 50 Kg.
* Refusal to participate in the study (absence of informed consent).
* Patient with chronic kidney disease on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Analyze filter/system useful life | 72 hours per filter
  Evaluate the duration of the continuous hemodiafiltration filter according to changes in blood flow

SECONDARY OUTCOMES:
Examine the system pressures | 72 hours per filter
  Assess changes in system pressures during the 2 blood flows (transmembrane pressure, filter pressure and access pressure)
Assess filtration fraction variation | 72 hours per filter
  Assess filtration fraction variation during the 2 blood flows
Electrolytic control - Potassium | 72 hours per filter (dosage every 12 hours according to protocol)
  Assess changes in potassium (changes from baseline)
Electrolytic control - Sodium | 72 hours per filter (dosage every 12 hours according to protocol)
  Assess changes in sodium (changes from baseline)
Acid-base balance - blood pH | 72 hours per filter (venous blood gas analysis every 12 hours)
  Assess changes in blood pH during the 2 blood flows (changes from baseline)
Acid-base balance - sodium bicarbonate | 72 hours per filter (venous blood gas analysis every 12 hours)
  Assess changes in sodium bicarbonate during the 2 blood flows (changes from baseline)
Acid-base balance - base excess | 72 hours per filter (venous blood gas analysis every 12 hours)
  Assess changes in base excess during the 2 blood flows (changes from baseline)
Mortality of the cohort | 30, 60 and 90 days
  Assess the overall mortality of the cohort in 30, 60 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Lucas T Avila Neto, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelite Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kellum JA, Romagnani P, Ashuntantang G, Ronco C, Zarbock A, Anders HJ. Acute kidney injury. Nat Rev Dis Primers. 2021 Jul 15;7(1):52. doi: 10.1038/s41572-021-00284-z. PMID 34267223
- [Background] Fuhrman DY, Kellum JA. Acute Kidney Injury in the Intensive Care Unit: Advances in the Identification, Classification, and Treatment of a Multifactorial Syndrome. Crit Care Clin. 2021 Apr;37(2):xiii-xv. doi: 10.1016/j.ccc.2021.01.001. Epub 2021 Feb 13. No abstract available. PMID 33752867
- [Background] Bellomo R, Baldwin I, Ronco C, Kellum JA. ICU-Based Renal Replacement Therapy. Crit Care Med. 2021 Mar 1;49(3):406-418. doi: 10.1097/CCM.0000000000004831. No abstract available. PMID 33555775
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Khadzhynov D, Schelter C, Lieker I, Mika A, Staeck O, Neumayer HH, Peters H, Slowinski T. Incidence and outcome of metabolic disarrangements consistent with citrate accumulation in critically ill patients undergoing continuous venovenous hemodialysis with regional citrate anticoagulation. J Crit Care. 2014 Apr;29(2):265-71. doi: 10.1016/j.jcrc.2013.10.015. Epub 2013 Nov 11. PMID 24360392
- [Background] Gattas DJ, Rajbhandari D, Bradford C, Buhr H, Lo S, Bellomo R. A Randomized Controlled Trial of Regional Citrate Versus Regional Heparin Anticoagulation for Continuous Renal Replacement Therapy in Critically Ill Adults. Crit Care Med. 2015 Aug;43(8):1622-9. doi: 10.1097/CCM.0000000000001004. PMID 25853591
- [Background] Stucker F, Ponte B, Tataw J, Martin PY, Wozniak H, Pugin J, Saudan P. Efficacy and safety of citrate-based anticoagulation compared to heparin in patients with acute kidney injury requiring continuous renal replacement therapy: a randomized controlled trial. Crit Care. 2015 Mar 18;19(1):91. doi: 10.1186/s13054-015-0822-z. PMID 25881975
- [Background] Meersch M, Kullmar M, Wempe C, Kindgen-Milles D, Kluge S, Slowinski T, Marx G, Gerss J, Zarbock A; SepNet Critical Care Trials Group. Regional citrate versus systemic heparin anticoagulation for continuous renal replacement therapy in critically ill patients with acute kidney injury (RICH) trial: study protocol for a multicentre, randomised controlled trial. BMJ Open. 2019 Jan 21;9(1):e024411. doi: 10.1136/bmjopen-2018-024411. PMID 30670518
- [Background] Zarbock A, Kullmar M, Kindgen-Milles D, Wempe C, Gerss J, Brandenburger T, Dimski T, Tyczynski B, Jahn M, Mulling N, Mehrlander M, Rosenberger P, Marx G, Simon TP, Jaschinski U, Deetjen P, Putensen C, Schewe JC, Kluge S, Jarczak D, Slowinski T, Bodenstein M, Meybohm P, Wirtz S, Moerer O, Kortgen A, Simon P, Bagshaw SM, Kellum JA, Meersch M; RICH Investigators and the Sepnet Trial Group. Effect of Regional Citrate Anticoagulation vs Systemic Heparin Anticoagulation During Continuous Kidney Replacement Therapy on Dialysis Filter Life Span and Mortality Among Critically Ill Patients With Acute Kidney Injury: A Randomized Clinical Trial. JAMA. 2020 Oct 27;324(16):1629-1639. doi: 10.1001/jama.2020.18618. PMID 33095849
- [Background] Kramer L, Bauer E, Joukhadar C, Strobl W, Gendo A, Madl C, Gangl A. Citrate pharmacokinetics and metabolism in cirrhotic and noncirrhotic critically ill patients. Crit Care Med. 2003 Oct;31(10):2450-5. doi: 10.1097/01.CCM.0000084871.76568.E6. PMID 14530750
- [Background] Bauer E, Derfler K, Joukhadar C, Druml W. Citrate kinetics in patients receiving long-term hemodialysis therapy. Am J Kidney Dis. 2005 Nov;46(5):903-7. doi: 10.1053/j.ajkd.2005.07.041. PMID 16253731
- [Background] Yu W, Zhuang F, Ma S, Fan Q, Zhu M, Ding F. Optimized Calcium Supplementation Approach for Regional Citrate Anticoagulation. Nephron. 2019;141(2):119-127. doi: 10.1159/000494693. Epub 2018 Nov 16. PMID 30448847
- [Background] Schneider AG, Journois D, Rimmele T. Complications of regional citrate anticoagulation: accumulation or overload? Crit Care. 2017 Nov 19;21(1):281. doi: 10.1186/s13054-017-1880-1. PMID 29151020
- [Background] AYRES, M., AYRES Jr, M., AYRES, D. L., SANTOS, A. A. S. Bioestat 5.3 aplicações estatísticas nas áreas das ciências biológicas e médicas. Belém: IDSM, 2007.364p.